CLINICAL TRIAL: NCT00216034
Title: Randomized Multicenter Controlled Phase III Study of Postoperative Adjuvant Therapy for Stage II/IIIA Gastric Cancer Using TS-1 Alone or TS-1+PSK Combined Therapy
Brief Title: Randomized Controlled Study of Postoperative Adjuvant Therapy for Gastric Cancer Using TS-1 or TS-1+PSK
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hokuriku-Kinki Immunochemotherapy Study Group (Other)
Responsible Party: Principal Investigator, Takashi Fujimura, Assistant Professor of Gastroenterologic Surgery, Kanazawa University Hospital, Hokuriku-Kinki Immunochemotherapy Study Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HKIT-GC
Record Dates: First submitted 2005-09-18; First posted 2005-09-22 (Estimated); Last update posted 2016-06-07 (Estimated); Status verified 2016-06

CONDITIONS: Gastric Cancer
Keywords: Gastric Cancer; TS-1; PSK; Disease-free survival; Overall survival
MeSH Terms: conditions — Stomach Neoplasms | interventions — titanium silicide; polysaccharide-K

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): TS-1 Group: The group treated with TS-1 mono-therapy
  Interventions: Drug: Tegafur-gimeracil-oteracil potassium (TS-1)
- 2 (Experimental): TS-1+PSK Group: The group treated with combination therapy using TS-1 and PSK
  Interventions: Drug: Tegafur-gimeracil-oteracil potassium (TS-1); Drug: Krestin (PSK)

INTERVENTIONS:
Drug: Tegafur-gimeracil-oteracil potassium (TS-1) — From 4-8 weeks after surgery to 27-31 weeks after surgery, 80 mg/m2, PO from day 1 to day 14 of each 21 day cycle. Number of Cycles: 8 From 28-32 weeks after surgery to 53-57 weeks after surgery, 80 mg/m2, PO from day 1 to day 14 of each 28 day cycle. Number of Cycles: 7
  Other Names: TS-1
Drug: Krestin (PSK) — From 4-8 weeks after surgery to 53-57 weeks after surgery, 3 g/day, PO every day
  Other Names: PSK
  Arms: 2

SUMMARY:
A randomized controlled study is conducted on patients with resected gastric cancer assigned to postoperative adjuvant therapy of TS-1 alone or PSK combined with TS-1, with the objective to examine or validate the outcome, QOL and prognostic factors (host and tumor factors), and explore the factors enhancing the antitumor effect of TS-1.

DETAILED DESCRIPTION:
The 5-year survival after gastric cancer surgery remains poor as the cancer advances to stages II, IIIA, IIIB and IV. Tegafur-gimeracil-oteracil potassium (TS-1) is used as the first line treatment for advanced and recurrent gastric cancer. But TS-1 is accompanied by an adverse drug reaction of bone marrow suppression that is not readily seen in conventional oral fluoropyrimidines. Among randomized controlled trials on postoperative adjuvant chemotherapy for gastric cancer, the beneficial results of survival rates using Krestin (PSK) in combination with chemotherapy have been reported. With the objective to enhance the antitumor effect of TS-1 and to improve the QOL of patients, we have planned to validate the clinical significance of combined PSK and TS-1 therapy as postoperative adjuvant therapy for gastric cancer, using in principle the TS-1 regimen of 2-week dosing 1-week off for 6 months followed by 2-week dosing 2-week off for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with microscopic stage II or IIIA resectable gastric cancer
* Patients who have not received preoperative cancer therapy (radiotherapy, chemotherapy or immunotherapy)
* Patients with serum immunosuppressive acidic protein (IAP) measured within 2 weeks before surgery
* Patients with no metachronous or synchronous multiple cancer
* Patients without severe impairment of renal, hepatic and bone marrow functions
* Patients who are judged to be capable of tolerating surgery
* Patients with preoperative performance status 0 to 2
* Patients with no serious concurrent complications (such as bone marrow suppression, diarrhea and infection)
* Patients who are judged to be capable of tolerating this treatment, and who have given written informed consent to participate in this study

Exclusion Criteria:

* Patients with fresh hemorrhage from the gastrointestinal tract
* Patients with retention of body fluid necessitating treatment
* Patients with infection, intestinal palsy or intestinal occlusion
* Patients who are pregnant or hope to become pregnant during the study period
* Patients with diabetes treated by continuous use of insulin or showing poor glycemic control
* Patients with a history of ischemic heart disease
* Patients with concurrent psychiatric disease or psychotic symptoms, and judged to have difficulties participating in the study
* Patients receiving continuous administration of steroids
* Patients who have experienced serious drug allergy in the past
* Others, patients judged by the investigator or subinvestigator to be inappropriate as subject

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2005-03; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Time of recurrence (calculation of 3-year disease-free survival and overall survival rates) | Five years after surgery

SECONDARY OUTCOMES:
Relations of survival rate with compliance, postoperative complication, QOL, adverse events, recurrence status, and expression of immune or tumor markers | Five years after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Koichi Miwa, MD, PhD, Study Chair — Hokuriku-Kinki Immunochemotherapy Study Group
Locations (42):
- Japan (42):
  - Fukui Cardio Vascular Center, Fukui-shi, Fukui
  - Fukui General Hospital, Fukui-shi, Fukui
  - Fukui Saiseikai Hospital, Fukui-shi, Fukui
  - University of Fukui Hospital, Iijima, Fukui
  - National Hospital Organization Fukui Hospital, Tsuruga, Fukui
  - Gifu Municipal Hospital, Gifu, Gifu
  - Gifu Prefectural General Medical Center, Gifu, Gifu
  - Gifu University Hospital, Gifu, Gifu
  - Shakaihoken Kobe Central Hospital, Kobe, Hyōgo
  - Public Central Hospital of Matto Ishikawa, Hakusan, Ishikawa-ken
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Ishikawa Prefectural Central Hospital, Kanazawa, Ishikawa-ken
  - Kanazawa Redcross Hospital, Kanazawa, Ishikawa-ken
  - Kanazawa Medical University Hospital, Mukai-awagasaki, Ishikawa-ken
  - Fukuchiyama City Hospital, Fukuchiyama, Kyoto
  - Kyoto Ohashi General Hospital, Fushimi, Kyoto
  - Houyu hospital, Jōyō, Kyoto
  - Saiseikai Kyoto Hospital, Kōtari, Kyoto
  - University Hospital, Kyoto Prefectural University of Medicine, Kyoto, Kyoto
  - Nishijin Hospital, Kyoto, Kyoto
  - Kyoto First Red Cross Hospital, Kyoto, Kyoto
  - National Hospital Organization Maizuru Medical Center, Maizuru, Kyoto
  - Nantan General Hospital, Nantan, Kyoto
  - Rokujizo Hospital, Uji, Kyoto
  - Second Okamoto General Hospital, Uji, Kyoto
  - Kyoto Prefectural Yosanoumi Hospital, Yotsutsuji, Kyoto
  - Marutamachi Hospital, Nishinokyokurumazaka-cho, Nakagyou-ku Kyoto
  - Nara City Hospital, Nara, Nara
  - Matsushita Memorial Hospital, Moriguchi, Osaka
  - Osaka Railway hospital, Osaka, Osaka
  - Midorigaoka Hospital, Takatsuki, Osaka
  - Osaka City University Hospital, Kembuchi, Osaka Abeno-ku
  - Sumitomo Hospital, Nakanoshima, Osaka Kita-ku
  - Shiga University of Medical Science Hospital, Ōtsu, Shiga
  - Saiseikai Shigaken Hospital, Rittō, Shiga
  - Shimane University Hospital, Izumo, Shimane
  - Saiseikai Takaoka Hospital, Takaoka, Toyama
  - Kouseiren Takaoka Hoapital, Takaoka, Toyama
  - Toyama Prefectural Central Hospital, Toyama, Toyama
  - Toyama Rosai Hospital, Uozu, Toyama
  - Yatsuo General Hospital, Yatsuomachi-higashikumisaka, Toyama
  - Kitade Hospital, Gobou, Wakayama

REFERENCES:
- [Background] Nakazato H, Koike A, Saji S, Ogawa N, Sakamoto J. Efficacy of immunochemotherapy as adjuvant treatment after curative resection of gastric cancer. Study Group of Immunochemotherapy with PSK for Gastric Cancer. Lancet. 1994 May 7;343(8906):1122-6. doi: 10.1016/s0140-6736(94)90233-x. PMID 7910230
- [Derived] Ueda Y, Fujimura T, Kinami S, Hirono Y, Yamaguchi A, Naitoh H, Tani T, Kaji M, Yamagishi H, Miwa K; Hokuriku-Kinki Immunochemo-Therapy Study Group-Gastric Cancer (HKIT-GC). A randomized phase III trial of postoperative adjuvant therapy with S-1 alone versus S-1 plus PSK for stage II/IIIA gastric cancer: Hokuriku-Kinki Immunochemo-Therapy Study Group-Gastric Cancer (HKIT-GC). Jpn J Clin Oncol. 2006 Aug;36(8):519-22. doi: 10.1093/jjco/hyl048. Epub 2006 Jun 27. PMID 16803844